CLINICAL TRIAL: NCT00083811
Title: HYPGENE-Genetics Fitness Obesity & Risk of Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1252; R01HL069870 (NIH)
Record Dates: First submitted 2004-06-02; First posted 2004-06-04 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2008-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity

SUMMARY:
To investigate the role of genetics in cardiorespiratory fitness, obesity, and risk of hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension is a multifactorial disease with genetic and environmental factors contributing to the disease process. HYPGENE will investigate gene-fitness and gene-obesity interactions that relate to the development of hypertension during adulthood. The study uses the cohort of the Aerobics Center Longitudinal Study (ACLS) at the Cooper Clinic.

DESIGN NARRATIVE:

The HYPGENE Study is a collaborative effort between the Pennington Biomedical Research Center, the Cooper Institute, and Washington University in St. Louis. The aim of the study is to investigate the contributions of DNA sequence variation in candidate genes as well as their interactions with cardiorespiratory fitness and obesity to the risk of hypertension in participants of the Aerobics Center Longitudinal Study (ACLS). In the first phase (as of 12/01/03), a group of 1000 subjects, who were normotensive and free of cardiovascular disease and diabetes at the time of their first preventive medical examination (from 01/1987 to 02/2001) will be selected from the ACLS cohort. Half of these subjects (n=500) developed hypertension during the follow-up period (duration 2 to 16 years), whereas the other half remained normotensive. In the second phase (from 12/03 to 11/05), the sample size will be increased to 1500 subjects (750 cases and 750 controls). Cases are defined as individuals who were normotensive at baseline but developed essential hypertension during follow-up. Comparison individuals are those who also were normotensive at baseline and remained normotensive during follow-up. The ascertainment of the case-control status will be done during the subjects' return visits to the Cooper Clinic. A panel of biallelic single nucleotide polymorphisms in candidate gene loci will be typed. The candidate genes are selected based on their putative roles in the physiological pathways pertaining to the regulation of blood pressure by fitness and obesity, or on evidence of linkages and associations in previous studies. The candidates include endothelial factors contributing to vasodilation and vasoconstriction, beta-adrenergic receptors and their kinases, which mediate the effects of autonomic nervous system on cardiac function and vascular tone, the renin angiotensin system, and signaling molecules that mediate the effects of laminar shear stress on vascular wall enzyme activity and gene expression. Logistic regression modeling and classification and regression trees methodology will be used to analyze the contribution of genotype, fitness level and obesity, as well as their interactions, to the risk of hypertension. The HYPGENE study will produce novel data on the effects of genetic factors in the presence of either high or low cardiorespiratory fitness level or obesity or normal body weight on the development of hypertension. These data could ultimately lead to more efficient use of physical activity and body weight control in the primary and secondary prevention of hypertension.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tuomo Rankinen — Pennington Biomedical Research Center